CLINICAL TRIAL: NCT06679465
Title: Evaluating the Impact of Single Dose Tiotropium on Allergen-induced Early Asthmatic Response
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Brianne Philipenko, MD FRCPC, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 5080
Record Dates: First submitted 2024-10-25; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Asthma Bronchiale
Keywords: asthma; Tiotropium; Early asthmatic response
MeSH Terms: conditions — Asthma | interventions — Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tiotropium treatment (Experimental): 2 puffs tiotropium
  Interventions: Drug: Tiotropium (Spiriva®)
- Placebo (Placebo Comparator): 2 puffs placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tiotropium (Spiriva®) — 2 puffs tiotropium prior to allergen challenge
  Arms: Tiotropium treatment
Drug: Placebo — 2 puffs placebo
  Arms: Placebo

SUMMARY:
Evaluate single dose (2 x 2.5mcg/puff; total dose 5mcg) effect of tiotropium administered 30 minutes prior to allergen challenge on allergen-induced EAR assessed as the maximal % fall in FEV1 after allergen inhalation compared to that of single dose (two puffs) matched placebo administered 30 minutes prior to allergen challenge.

ELIGIBILITY:
Inclusion Criteria:

* age (years) at least 18 years
* no confounding health issue (i.e. no health conditions, other than asthma, that would put the participant at risk or affect data integrity as determined by the principal investigator)
* baseline FEV1 ≥ 65% of predicted normal at Visit 1
* evidence of atopy to an allergen suitable for inhalation challenge following skin prick testing such as house dust mite, grass, cat or horse
* fall in FEV1 of ≥ 20% at a dose of methacholine ≤ 600mcg (methacholine PD20) at Visit 1
* positive response to allergen inhalation challenge (fall in FEV1 of ≥ 15% after inhalation of allergen at a dilution 1:32 or more dillute.
* absence of respiratory infection for at least 4 weeks prior to Visit 1
* absence of significant worsening of asthma that requires health care intervention or prolonged change in medication due to allergen exposure (or other trigger) for at least 4 weeks prior to Visit 1
* women of child-bearing potential shall not be pregnant or lactating
* non-smoker (cigarettes, vaping); ex-smoker with <10 pack year history allowed; cannabis use will be evaluated on a case-by-case basis
* if on as needed budesonide/formoterol therapy, no reported use within 3 weeks prior to allergen challenge

Exclusion Criteria:

* Smoker >10 pack year history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Early asthmatic response | 2 hours post-allergen challenge
  Evaluate single dose (2 x 2.5mcg/puff; total dose 5mcg) effect of tiotropium administered 30 minutes prior to allergen challenge on allergen-induced EAR assessed as the maximal % fall in FEV1 after allergen inhalation compared to that of single dose (two puffs) matched placebo administered 30 minutes prior to allergen challenge.

SECONDARY OUTCOMES:
Inflammatory response | Five hours post-allergen challenge
  1. Evaluate effect of single dose tiotropium versus single dose matched placebo on airway inflammation five hours after allergen challenge through analyses of sputum eosinophil counts, and cytokine analysis including IL-4, 5, 13 and TSLP.
FEV1 | 30 minutes
  2. Evaluate bronchodilating effect of single dose tiotropium versus placebo on baseline lung function by comparing maximal FEV1 pre versus 30 minutes post treatment (i.e. prior to allergen challenge).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No